CLINICAL TRIAL: NCT00021892
Title: Ventricular Matrix Remodeling: Correlates and Prognosis
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 973; R01HL067288 (NIH)
Record Dates: First submitted 2001-08-10; First posted 2001-08-10 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Heart Diseases; Heart Failure, Congestive; Cardiovascular Diseases; Heart Failure
MeSH Terms: conditions — Heart Diseases; Heart Failure; Cardiovascular Diseases

SUMMARY:
To assess the diagnostic and prognostic usefulness of serum markers of left ventricular remodeling for predicting congestive heart failure.

DETAILED DESCRIPTION:
BACKGROUND:

Recent studies have established that cardiac extracellular matrix (ECM) remodeling is a major determinant of pathologic left ventricular hypertrophy (LVH) and progressive left ventricular dilatation, and as a result, contributes to the development of left ventricular dysfunction and overt congestive heart failure (CHF). The recent development of reliable serologic assays for procollagen peptides, metalloproteinases (MMP) and their tissue inhibitors (TIMP), and cytokines permits the in vivo assessment of LV ECM remodeling, and raises the possibility of expanding the utility of these markers 'from the bench to the bedside.' Prior studies of ECM biomarkers in congestive heart failure have been limited to cross-sectional investigations of small samples of highly selected patients with advanced disease. The fundamental question whether serum markers of ECM remodeling are important correlates of left ventricular dilatation or left ventricular hypertrophy, or are independent predictors of incident congestive heart failure in the community remains unanswered.

DESIGN NARRATIVE:

The aims of the study are to: determine the relationships between serum markers of ECM remodeling and traditional congestive heart failure risk factors; analyze the cross-sectional relations between markers of ECM remodeling and echocardiographic left ventricular hypertrophy and left ventricular dilatation, Doppler indices of left ventricular filling and serum natriuretic peptides; investigate prospectively the relationships between ECM remodeling markers and progressive left ventricular dilatation and left ventricular hypertrophy and congestive heart failure incidence, adjusting for standard risk factors. Stored samples from the Framingham Offspring and Omni cohorts will be used. Participants at the extremes of the joint distributions of left ventricular wall thickness and left ventricular internal dimension from echocardiograms performed at earlier Framingham exams will be sampled.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-06; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vasan Ramachandran — Boston University

REFERENCES:
- [Background] Sundstrom J, Evans JC, Benjamin EJ, Levy D, Larson MG, Sawyer DB, Siwik DA, Colucci WS, Sutherland P, Wilson PW, Vasan RS. Relations of plasma matrix metalloproteinase-9 to clinical cardiovascular risk factors and echocardiographic left ventricular measures: the Framingham Heart Study. Circulation. 2004 Jun 15;109(23):2850-6. doi: 10.1161/01.CIR.0000129318.79570.84. Epub 2004 Jun 1. PMID 15173025
- [Background] Kathiresan S, Larson MG, Benjamin EJ, Corey D, Murabito JM, Fox CS, Wilson PW, Rifai N, Meigs JB, Ricken G, Lifton RP, Levy D, Vasan RS. Clinical and genetic correlates of serum aldosterone in the community: the Framingham Heart Study. Am J Hypertens. 2005 May;18(5 Pt 1):657-65. doi: 10.1016/j.amjhyper.2004.12.005. PMID 15882548
- [Background] Dhingra R, Ho Nam B, Benjamin EJ, Wang TJ, Larson MG, D'Agostino RB Sr, Levy D, Vasan RS. Cross-sectional relations of electrocardiographic QRS duration to left ventricular dimensions: the Framingham Heart Study. J Am Coll Cardiol. 2005 Mar 1;45(5):685-9. doi: 10.1016/j.jacc.2004.11.046. PMID 15734611